CLINICAL TRIAL: NCT05140928
Title: The Effect of Maternal Dadiah (Minangkabau Yogurt) Supplementation During Pregnancy on Child Growth, Gut Microbiota Proportion and the Level of Secretory Immunoglobulin A, in West Sumatra: A Randomised Clinical Trial
Brief Title: The Effect of Maternal Dadiah Supplementation During Pregnancy on Child Growth and Gastrointestinal Health Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Andalas University (Other)
Collaborators: Indonesia University (Other)
Responsible Party: Principal Investigator, Zuhrah Taufiqa, Principal Investigator, Andalas University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: III/UN.16.2/KEP-FK/2020; NKB3239/UN2.RST/HKP.05.00/2020 (Other Grant/Funding Number: PUTI Grant by Universitas Indonesia)
Record Dates: First submitted 2021-11-18; First posted 2021-12-02 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-12

CONDITIONS: Gastrointestinal Microbiome; Immunoglobulin A; Growth; Stunting, Nutritional
Keywords: dadiah; local yogurt; Minangkabau yogurt; pregnant women; dietary supplement; gut microbiota; immunoglobulin A; gastrointestinal health; fermented dairy product; lactic acid bacteria; child growth; probiotic
MeSH Terms: conditions — Growth Disorders

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to two groups; the intervention group that received dadiah pudding and the control group that received pudding without dadiah in parallel for the duration of the study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dadiah Pudding (Active Comparator): The mother received 1 cup or 100 g dadiah pudding containing 75-gram dadiah which provide ±260 kcal energy, 6.12g protein, 23.31g fat, 6.49g carbohydrate, and 6.1x 109 CFU/ml lactic acid bacteria.
  Interventions: Other: Dadiah Pudding
- Pudding without dadiah (Placebo Comparator): The mother received 1 cup or 100 g pudding without dadiah containing ±75 kcal energy, 0.3g protein, 0.45 g fat, and 16.2g carbohydrate.
  Interventions: Other: Pudding without Dadiah

INTERVENTIONS:
Other: Dadiah Pudding — Supplementation of Dadiah Pudding to pregnant women. One cup a day for 18-26 weeks of pregnancy
  Other Names: Minangkabau Yogurt Pudding
  Arms: Dadiah Pudding
Other: Pudding without Dadiah — Supplementation of Milk Pudding without dadiah to pregnant women. One cup a day for 18-26 weeks of pregnancy
  Other Names: Milk Pudding
  Arms: Pudding without dadiah

SUMMARY:
The aim of our study is to assess the effect of giving dadiah as a supplement to pregnant women on improving the growth and digestive health of children.

DETAILED DESCRIPTION:
The study was carried out on pregnant women in four Public Health Center (PHC) areas in Padang Panjang, West Sumatra, Indonesia. They were screened for inclusion and exclusion criteria. Once eligibility was confirmed, pregnant women were randomly allocated to intervention or control groups. The details of the study protocol were explained, and voluntary written consent was obtained.

General information about the mother was collected and a general physical examination was assessed. The intervention started at about 10-20 weeks of gestation and continued until just before the time of delivery. Subjects took the study supplements concurrently with the government's dietary supplementation program. In each home visit, the remaining supplements from the previous visit were counted and documented in the pudding checklist form. Details of symptoms or illnesses during consumption of dadiah pudding will be reported either by participants directly contacting field officers, study staff, or during weekly visits and will be recorded and documented in the case report form. In the third trimester, subjects received healthy food, breastfeeding practices, and child development education to support mothers in maintaining their nutritional status, preparing exclusive breastfeeding, and optimizing child development.

Healthy babies born to mothers will be the focus of this study and followed up until the age of three months to assess their growth. The information includes the baby's health history after birth, anthropometric measurements, nutritional intake, and breastfeeding practices which are measured repeatedly in the first, second, and third months. The collection of breast milk and baby feces is carried out in the first week and third month after the baby is born.

The sample size was calculated taking into account all outcome variables including the proportion of gut microbiota, levels of IgA secretion in breast milk and infant feces, and child growth, with the independent variable being maternal supplementation during pregnancy.

Data quality assurance is carried out through training starting from the period of data collection and supervision during and after data collection, including the data analysis process. This included training for enumerators, subjects and using a validated questionnaire for a group of subjects representing similar characteristics for this study. Data input and cleaning process will use excel and SPSS while for food intake data using NutriSurvey 2007. Data entry will be carried out by data collection officers after data collection. The data cleaning process includes removing outliers and regrouping multiple results that have similar meanings. The data will be interpreted as mean ± standard deviation if the data is normally distributed and the median (min-max) if the data is not normally distributed. Statistical analysis using SPSS 20 and data will be analyzed using univariate and bivariate analysis. Univariate analysis is used to describe characteristics and socio-demographics, medical history, pregnancy, and obstetric profiles of pregnant women. Numerical variables between groups will be analyzed using an Independent sample t-test if the data has normal distribution or the Mann Whitney test if the data distribution is not normal. Categorical variables between groups will be analyzed using Chi-square or Fisher test. Differences between birth and 3 months old follow up will be analyzed using Dependent t-tests if the data distribution has normal distribution or Wilcoxon test if the data distribution is not normal.

ELIGIBILITY:
Inclusion Criteria:

* Women with10-20 weeks gestation
* Women give voluntary informed consent
* Women willing to give exclusive breastfeeding
* Women live in an area under study, registered, and visit antenatal care at targeted public health centers
* Women plan to deliver babies in the area under study

Exclusion Criteria:

* Women having a medical history of HIV/AIDS, TBC, Hepatitis B.
* Women with multiple pregnancies
* Women having obesity, and/or another high-risk pregnancy (hypertension, preeclampsia, diabetes, bleeding history)
* Received antibiotic treatment or intentionally consumes probiotic products during the preceding 4 weeks. (If the subject was on antibiotics before the beginning of the study or probiotics, a washout period of 2 weeks is required.)

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2020-08-20 (Actual); Primary Completion 2021-09-09 (Actual); Study Completion 2021-09-09 (Actual)

PRIMARY OUTCOMES:
Infant fecal gut microbiota proportion | three months
  Relative difference of non-pathogen and pathogen to total bacteria in infant fecal sample
Breast milk gut microbiota proportion | three months
  Relative difference of non-pathogen and pathogen to total bacteria in infant fecal sample
Level of infant fecal secretory Immunoglobulin A | three months
  Concentration of secretory Immunoglobulin A in infant fecal sample
Level of breastmilk secretory Immunoglobulin A | three months
  Concentration of secretory Immunoglobulin A in breastmilk sample

SECONDARY OUTCOMES:
Weight increment | three months
  Change in body's relative mass of the child measured by subtract child weight at three months old to child weight in the first week
Length increment | three months
  Change in distance from the bottom of the feet to the top of the head in child's body fully extended and feet flexed measured by subtract child weight at three months old to child length in the first week
Head circumferences increment | three months
  Change in the circumference of the distance from above the eyebrows and ears and around the back of the head as a parameter in evaluate nutritional status measured by subtract child head circumference at three months old to child head circumference in the first week

CONTACTS AND LOCATIONS:
Overall Officials: Zuhrah Taufiqa, MD, Study Director — Indonesia University
Locations (1):
- Zuhrah Taufiqa, Padang, West Sumatra, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rinita Amelia, Koshy Philip, Yudha Endra Pratama EP. Characterization and probiotic potential of lactic acid bacteria isolated from dadiah sampled in West Sumatra. Food Sci Technol. 2020
- [Background] Taufiqa Z, Chandra DN, Helmizar H, Lipoeto NI, Hegar B. Micronutrient Content and Total Lactic Acid Bacteria of Dadiah Pudding as Food Supplementation for Pregnant Women. 2021;9:1149-55
- [Result] Collado MC, Surono IS, Meriluoto J, Salminen S. Potential probiotic characteristics of Lactobacillus and Enterococcus strains isolated from traditional dadih fermented milk against pathogen intestinal colonization. J Food Prot. 2007 Mar;70(3):700-5. doi: 10.4315/0362-028x-70.3.700. PMID 17388062
- [Result] Surono IS. Traditional Indonesian dairy foods. Asia Pac J Clin Nutr. 2015;24 Suppl 1:S26-30. doi: 10.6133/apjcn.2015.24.s1.05. PMID 26715081
- [Result] Surono IS, Martono PD, Kameo S, Suradji EW, Koyama H. Effect of probiotic L. plantarum IS-10506 and zinc supplementation on humoral immune response and zinc status of Indonesian pre-school children. J Trace Elem Med Biol. 2014 Oct;28(4):465-9. doi: 10.1016/j.jtemb.2014.07.009. Epub 2014 Aug 2. PMID 25183688
- [Result] Mantaring J, Benyacoub J, Destura R, Pecquet S, Vidal K, Volger S, Guinto V. Effect of maternal supplement beverage with and without probiotics during pregnancy and lactation on maternal and infant health: a randomized controlled trial in the Philippines. BMC Pregnancy Childbirth. 2018 May 31;18(1):193. doi: 10.1186/s12884-018-1828-8. PMID 29855271
- [Result] Robertson RC. The Gut Microbiome in Child Malnutrition. Nestle Nutr Inst Workshop Ser. 2020;93:133-144. doi: 10.1159/000503352. Epub 2020 Jan 28. PMID 31991429
- [Result] Swartwout B, Luo XM. Implications of Probiotics on the Maternal-Neonatal Interface: Gut Microbiota, Immunomodulation, and Autoimmunity. Front Immunol. 2018 Dec 3;9:2840. doi: 10.3389/fimmu.2018.02840. eCollection 2018. PMID 30559747
- [Result] Chen Y, Li Z, Tye KD, Luo H, Tang X, Liao Y, Wang D, Zhou J, Yang P, Li Y, Su Y, Xiao X. Probiotic Supplementation During Human Pregnancy Affects the Gut Microbiota and Immune Status. Front Cell Infect Microbiol. 2019 Jul 16;9:254. doi: 10.3389/fcimb.2019.00254. eCollection 2019. PMID 31380297
- [Result] Baldassarre ME, Di Mauro A, Mastromarino P, Fanelli M, Martinelli D, Urbano F, Capobianco D, Laforgia N. Administration of a Multi-Strain Probiotic Product to Women in the Perinatal Period Differentially Affects the Breast Milk Cytokine Profile and May Have Beneficial Effects on Neonatal Gastrointestinal Functional Symptoms. A Randomized Clinical Trial. Nutrients. 2016 Oct 27;8(11):677. doi: 10.3390/nu8110677. PMID 27801789
- [Result] Prakoeswa CRS, Herwanto N, Prameswari R, Astari L, Sawitri S, Hidayati AN, Indramaya DM, Kusumowidagdo ER, Surono IS. Lactobacillus plantarum IS-10506 supplementation reduced SCORAD in children with atopic dermatitis. Benef Microbes. 2017 Oct 13;8(5):833-840. doi: 10.3920/BM2017.0011. Epub 2017 Oct 12. PMID 29022387
- [Result] Hill C, Guarner F, Reid G, Gibson GR, Merenstein DJ, Pot B, Morelli L, Canani RB, Flint HJ, Salminen S, Calder PC, Sanders ME. Expert consensus document. The International Scientific Association for Probiotics and Prebiotics consensus statement on the scope and appropriate use of the term probiotic. Nat Rev Gastroenterol Hepatol. 2014 Aug;11(8):506-14. doi: 10.1038/nrgastro.2014.66. Epub 2014 Jun 10. PMID 24912386